CLINICAL TRIAL: NCT00553956
Title: Phase 1:Epidemiological Study of PTSD and Comorbid Disorders in Widows and Orphans Who Experienced the Rwandan Genocide Phase 2: A Randomized Controlled Clinical Trial With Orphans and Widows Who Experienced the Genocide Carried Out by Trained Local Psychologists -NET/IPT Versus Waiting List-
Brief Title: A Randomized Controlled Clinical Trial With Orphans and Widows Who Experienced the Rwandan Genocide
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Konstanz (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NET_IPT
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Posttraumatic Stress Disorder; Depression; Prolonged Grief Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Prolonged Grief Disorder | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Intervention group A treatment combination of Narrative Exposure Therapy and Interpersonal Psychotherapy (5 individual sessions NET in addition to 3 individual sessions IPT)
  Interventions: Behavioral: Narrative Exposure Therapy/Interpersonal Psychotherapy
- 2 (No Intervention): Waiting list control

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy/Interpersonal Psychotherapy — The experimental group will receive 5 weekly individual sessions of NET in addition to 3 weekly individual sessions of IPT.
  Arms: 1

SUMMARY:
In the framework of the epidemiological study, local psychologists are trained in Butare in carrying out diagnostic interviews with orphans and widows who experienced the Rwandan genocide. With the aid of standardized questionnaires they will assess trauma related symptoms as well as Prolonged Grief Disorder. Under the supervision of clinical experts from the University of Konstanz the local psychologists will carry out a randomized house to house survey (Phase 1).

As a second step, a controlled randomized clinical trial will be carried out. Local psychologists will be trained in applying Narrative Exposure Therapy and Interpersonal Psychotherapy. Genocide survivors that will be identified with a PTSD diagnosis will randomly be assigned to either the treatment condition or a waiting list. The treatment group will receive 5 individual sessions of NET in addition to 3 individual IPT sessions. Subsequent 3-months and 6-months post-tests will serve to evaluate the efficacy of this treatment module in alleviating trauma related symptoms and symptoms of prolonged grief. We expect a significant symptom reduction in the experimental group and no significant symptom reduction in the waiting list. After the 6-months post-test, the trained psychologists will train other psychologists in applying this treatment module under the supervision of clinical experts from the University of Konstanz. Afterwards, they will apply therapy to the victims from the waiting list.

A 12-months follow-up will serve to evaluate the long-term effect of the NET/IPT combination.

ELIGIBILITY:
Inclusion Criteria:

* widows and orphans
* confrontation of the Rwandan genocide
* clinical diagnosis of PTSD

Exclusion Criteria:

* mental retardation
* psychotic symptoms
* current drug or alcohol

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-08; Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Symptoms of PTSD, depression, prolonged grief disorder | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Schaal, Principal Investigator — University of Konstanz
Locations (1):
- Victims Voice, Butare, Province de Butare, Rwanda